CLINICAL TRIAL: NCT07399743
Title: Effects of Lower Body Positive Pressure Therapy Versus Alpha Lipoic Acid and Omega-3 Fatty Acids on Pain, Function, and Inflammation in Overweight Women With Knee Osteoarthritis: A Randomized Controlled Clinical Trial
Brief Title: Effects of Lower Body Positive Pressure Therapy Versus Alpha Lipoic Acid and Omega-3 Fatty Acids on Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Eman Said Sawan, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014233-49
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ALA tab 300 mg BID (Thioctacid) + PT (Active Comparator)
  Interventions: Drug: Alpha-Lipoic Acid (ALA)+PT
- Omega-3 cap 2000 mg BID (Limitless Omega) + PT (Active Comparator)
  Interventions: Drug: Omega-3 cap+ PT
- LBPP (AlterG 40-60% unload, 30 min 3×/week) + PT (Active Comparator)
  Interventions: Device: Lower body positive pressure therapy (LBPP)+PT
- PT (Active Comparator)
  Interventions: Device: Standard physical therapy (PT)

INTERVENTIONS:
Drug: Alpha-Lipoic Acid (ALA)+PT — Thioctacid 600+PT
  Arms: ALA tab 300 mg BID (Thioctacid) + PT
Drug: Omega-3 cap+ PT — Omega-3 cap 2000 mg BID (Limitless Omega) + PT
  Arms: Omega-3 cap 2000 mg BID (Limitless Omega) + PT
Device: Lower body positive pressure therapy (LBPP)+PT — LBPP: AlterG 40-60% unload, 30 min (3×/week) + PT
  Arms: LBPP (AlterG 40-60% unload, 30 min 3×/week) + PT
Device: Standard physical therapy (PT) — PT typically includes quadriceps strengthening, flexibility exercises, proprioceptive training, stationary cycling, and aquatic therapy
  Arms: PT

SUMMARY:
Here is a **concise, clear summary (~250 words / well under 5000 characters)** while preserving the key scientific points:

---

Knee osteoarthritis (KOA) is highly prevalent among overweight women, affecting more than 30% of those with BMI ≥25 kg/m². Excess body weight increases knee joint loading by 4-6 times per additional kilogram, accelerating cartilage degeneration, subchondral bone changes, and synovial inflammation. These alterations result in chronic pain, stiffness, functional limitation, and reduced quality of life, with obesity-related metabolic inflammation further worsening disease progression.

Standard physical therapy (PT) remains first-line treatment, yet provides only modest benefits, achieving approximately 15-20% WOMAC improvement at 12 weeks, while up to half of overweight patients continue to experience significant symptoms. Lower body positive pressure therapy (LBPP) via antigravity treadmill offers a biomechanical enhancement by unloading 40-80% of body weight, enabling pain-free gait training and reducing joint impact forces by up to 80%. Studies report 30-40% WOMAC improvement and better walking capacity compared with conventional PT.

Nevertheless, mechanical interventions alone do not address the inflammatory and oxidative mechanisms driving KOA. Alpha-lipoic acid (600 mg/day) and omega-3 fatty acids (1.5-2 g/day) provide targeted biochemical modulation, reducing pro-inflammatory cytokines, oxidative stress, and cartilage-degrading enzymes, with reported 25-35% functional improvement in clinical trials.

Despite the promise of both approaches, no randomized trial has directly compared adding LBPP versus combined ALA and omega-3 supplementation to standard PT in overweight women with KOA. This study aims to fill this gap by evaluating the relative effectiveness of biomechanical versus biochemical adjuncts to optimize management of KOA in this high-risk population.

ELIGIBILITY:
* Inclusion criteria

  1. Female participants aged between 20-45 years.
  2. Their BMI ranged between 20-25 kg/m².
  3. All had radiographic confirmation of mild to moderate knee osteoarthritis.
  4. Medical history recorded with no major prior injuries or surgeries affecting outcomes.
  5. Participants reported knee pain, functional limitation, and activity-related symptoms.
  6. Radiographic grading confirmed as Kellgren-Lawrence grade II or III.

Exclusion criteria:

1. No recent traumatic hip, knee, or ankle surgery within the past 6 months.
2. No severe knee OA (Kellgren-Lawrence grade 0 or 4).
3. No history of rheumatoid arthritis, chronic reactive arthritis, or psoriatic arthritis.
4. Free from conditions that limit safe study participation or adherence to protocol.
5. No neurological impairments affecting lower limb function.
6. No contraindications to exercise or physiotherapy (e.g., severe cardiovascular, respiratory, or metabolic conditions).
7. Not pregnant or planning pregnancy during the study.
8. Not involved in other clinical trials or conflicting interventions (e.g., intra-articular injections, surgery, or rehab programs).

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in VAS pain score (0-10 cm) | from baseline to 12 weeks
Change in WOMAC total score (0-96) | from baseline to 12 weeks

IPD SHARING:
Plan to Share IPD: No